CLINICAL TRIAL: NCT05516901
Title: Effect of Ultrasound Guided Erector Spinae Plane Block on Post-operative Pain and Diaphragmatic Dysfunction in Obese Patients Undergoing Epigastric Hernia Repair
Brief Title: Ultrasound Guided Erector Spinae Plane Block on Post-operative Pain and Diaphragmatic Dysfunction in Epigastric Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Asmaa Ragab Mohamed, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34579/3/21
Record Dates: First submitted 2022-08-20; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Epigastric Hernia Repair; Erector Spinae Plane Block; Post Operative Pain; Diaphragmatic Dysfunction
MeSH Terms: conditions — Pain, Postoperative | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Fifty obese patient BMI (30-40), aged (21-65) years ASA (ІΙ and ΙΙІ) and scheduled for elective Epigastric hernia repair were enrolled in the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Group allocation was done by sealed opaque envelope technique. All blocks were performed by the same anesthesiologist while the measurements were taken by another anesthesiologist who is blinded to the study groups and had no subsequent involvement in the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The erector spinae plane block group (Experimental): The erector spinae plane block group: Patients will receive general anesthesia plus bilateral ultrasound guided ESP block.
  Interventions: Procedure: The erector spinae plane block group
- Control group (Placebo Comparator): Control group (group І): Patients will receive general anesthesia alone.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: The erector spinae plane block group — The probe should then slowly be moved laterally until the transverse process is visible. The 100 mm, 25-gauge needle should be inserted using an in-plane approach in the cephalad to caudal direction and advanced under ultrasound guidance towards the transverse process; once the needle tip is below the erector spinae muscle, a small bolus of local anesthetic should be given. The erector spinae muscle should be visualized, separating from the transverse process. After aspiration the local anesthetic (20 ml of 0.25% bupivacaine was injected. Technique was repeated on the other side.
  Arms: The erector spinae plane block group
Procedure: Control group — Patients in this group will receive general anesthesia alone.
  Arms: Control group

SUMMARY:
The aim of this study is to assess the efficacy of ultrasound guided erector Spinae plane block on postoperative pain score and diaphragmatic dysfunction in obese patients undergoing Epigastric hernia repair.

DETAILED DESCRIPTION:
Ventral hernia repair is an operation associated with significant postoperative pain. There is a lot of modalities of pain control including regional anesthesia, intravenous opioids, and non-opioid analgesics. Regional anesthesia is often helpful in improving respiratory function and analgesia.

The dysfunction of the respiratory muscles, especially the diaphragm, caused by the upper abdominal surgery is a major cause of postoperative pulmonary complications, such as atelectasis and pneumonia. Sonografic evaluation of diaphragm is an accepted qualitative method of assessing diaphragmatic motion.

The erector spinae plane block is a paraspinal fascial plane block in which local anesthetic is administered between the erector spinae muscle and the transverse processes, blocking the dorsal and ventral rami of the thoracic and abdominal spinal nerves.

According to previous studies, erector spinae plane block provide lower postoperative pain score and decrease consumption of both postoperative and intraoperative analgesia for patients undergoing Epigastric hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Fifty obese patient BMI (30-40).
* Aged (21-65) years ASA (ІΙ and ΙΙІ)
* scheduled for elective Epigastric hernia repair

Exclusion Criteria:

* Patient refusal to continue the study.
* History of allergy to local anesthetics.
* Local infection at the site of the block.
* Patients with bleeding and coagulation disorders.
* Patients with renal, hepatic, cardiac dysfunction, or spine deformities.
* Patients with cognitive disorders.
* Patients with chronic pulmonary disease.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | 24 hours postoperatively.
  Post-operative pain will be assessed by Numeric Rating Scale at recovery room till 24 hours and if NRS˃3 morphine 3 mg will be given, total analgesics required will be recorded.
Diaphragmatic dysfunction by physiological parameter | 24 hours postoperatively.
  After recovery, patient laid in the supine position and diaphragm movements were recorded in the B-Mode and M-Mode. The probe was positioned between the midclavicular and anterior axillary lines, in the subcostal area, so that the ultrasound beam entered the posterior third of the right hemi diaphragm perpendicularly.
  After correct visualization of the right hemidiaphragm by B-mode, M-mode is used to display the motion of the diaphragm. At the end of normal expiration the patient was instructed to inhale as deeply as possible. A fixed point at the edge of the image on the screen and the diaphragm margin at maximal inspiration and again at maximal expiration served as reference points between which measurements were made, with the average of three values being taken for both maximal inspiration and maximal expiration

SECONDARY OUTCOMES:
Hypotension | 24 hours postoperatively
  defined as decrease blood pressure more than 20% of base line It was treated with rapid IV fluid infusion (100ml over 1 minutes) and bolus ephedrine 5-15 mg if needed.
Bradycardia | 24 hours postoperatively
  Bradycardia (heart rate less than 60 beats /minute) was treated with atropine 0.01mg/ kg

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt